CLINICAL TRIAL: NCT04385719
Title: An Open-label, Randomized, Single Intravenous Dosing Study to Investigate the Effect of Fixed-dose Combinations of Tenofovir/Lamivudine or Atazanavir/Ritonavir on the Pharmacokinetics of Remdesivir in Ugandan Healthy Volunteers
Brief Title: Drug-drug Interactions Between Remdesivir and Commonly Used Antiretroviral Therapy
Acronym: RemTLAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: University of Liverpool (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); University of Turin, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PK-24
Record Dates: First submitted 2020-03-29; First posted 2020-05-13 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Ebola; HIV/AIDS
Keywords: Ebola; HIV; Pharmacokinetics; Remdesivir; Drug Interactions
MeSH Terms: conditions — Hemorrhagic Fever, Ebola; Acquired Immunodeficiency Syndrome | interventions — remdesivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Study A Sequence 1 (Experimental): Single dose remdesivir 150mg IV on Day 1
  Wash out period Day 2-7
  TDF/3TC 300/300mg tablets OD from Day 8-14 single dose remdesivir 150mg IV on Day 14
  Interventions: Drug: Remdesivir
- Study A Sequence 2 (Experimental): TDF/3TC 300/300mg tablets OD from Day 1-7 single dose remdesivir 150mg IV on Day 7
  Wash out period Day 8-14
  Single dose remdesivir 150mg IV on Day 15
  Interventions: Drug: Remdesivir
- Study B (Experimental): TDF/3TC/ATV/r 300/300/300/100mg tablets OD from Day 1-7 single dose remdesivir 150mg IV infusion on Day 7
  Interventions: Drug: Remdesivir

INTERVENTIONS:
Drug: Remdesivir — Remdesivir (GS-5734) is a nucleoside analogue with in vitro activity against filoviruses EBOV, SUDV, BDBV and MARV, in addition to arenaviruses and coronaviruses
  Other Names: GS-5734

SUMMARY:
Ebola and HIV are found predominately in the same regions of the world and countries in sub-Saharan Africa are most affected by both diseases. For Ebola, no approved therapies exist. However, new investigational drugs are being evaluated to understand if they are effective against the Ebola virus. Remdesivir is an anti-Ebola investigational drug for the treatment of Ebola. Little is known about how the blood levels of remdesivir relate to how effective it is in patients with HIV taking antiretroviral therapy. This study will explore how commonly utilized ART (tenofovir/lamivudine and atazanavir/ritonavir) affect the drug levels of remdesivir.

DETAILED DESCRIPTION:
The study is designed as an open-label, randomized, fixed sequence, single intravenous dosing study to assess the effects of antiretrovirals on remdesivir pharmacokinetics.

The selection of healthy volunteers, as opposed to patients with HIV, avoids the greatest possible extent confounding factors, such as enzyme or transporter activity alteration in inflammatory states, concomitant medications potentially impacting drug disposition and other factors which are commonly present in a population of patients and cannot be easily eliminated.

Objectives:

Primary objective

1. To assess the safety and tolerability of single intravenous doses of remdesivir in adult healthy volunteers
2. To evaluate the intracellular pharmacokinetics of single dose intravenous remdesivir with or without co-administration of oral fixed-dose combination tenofovir/lamivudine with patients serving as their own controls

Secondary objectives

1. To evaluate the difference in plasma and intracellular pharmacokinetics of intravenous remdesivir among healthy volunteers receiving tenofovir/lamivudine versus healthy volunteers receiving tenofovir/lamivudine plus atazanavir/ritonavir tablets.
2. To generate a population pharmacokinetic model to describe inter-individual variability in intracellular pharmacokinetics of remdesivir

Exploratory objectives

1. To describe polymorphic variants of relevant kinases that activate TFV and explore possible consequences on remdesivir PK.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study.
2. Participants who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
3. Healthy men and women aged 18 to 55 years of age, and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
4. At screening, and all other visits, vital signs (systolic and diastolic blood pressure and pulse rate) will be assessed in the sitting position and again (when required) in the standing position. Sitting vital signs should be within the following ranges:

   I. axillary body temperature between 35.5-37.0 °C II. systolic blood pressure, 90-139 mmHg III. diastolic blood pressure, 50-89 mmHg IV. Pulse rate, 50-90 bpm. If pulse rate is between 40 and 50 bpm, the Investigator may decide to enroll the subject if he/she has history of athletic practice or other regular high cardio-vascular activity and ECG assessment is within normal range.

   Subjects should be excluded if their standing vital signs (relative to sitting) show findings which, in the opinion of the Investigator, are associated with clinical manifestation of postural hypotension (i.e. absence of any other cause). The Investigator should carefully consider enrolling subjects with either a > 20 mmHg decrease in systolic or a >10 mm Hg decrease in diastolic blood pressure, accompanied by a > 20 bpm increase in heart-rate (from sitting to standing).
5. Subjects must weigh at least 40 kg to participate in the study and must have a body mass index (BMI) within the range 18-30 Kg/m2. BMI= Body weight (kg) / [Height (m)]2
6. HIV antibody negative at screening.
7. Women of childbearing potential must be willing to use a highly effective contraception method (eg. IUD or hormonal contraceptive implant, complete abstinence (if genuinely followed)) or consistent use of a barrier method such as male or female condoms plus oral progestin contraceptives for the duration of the study. Non-surgically sterilized men must agree to abstain from sexual intercourse for the duration of the study or use condoms for contraception for the duration of the study.
8. Hemoglobin concentration equal or greater than 10 g/dL

Exclusion Criteria:

1. Significant disease affecting cardiac, respiratory, gastrointestinal or neurological symptoms which in the clinician's medical judgment could be worsened by participating in this study or the presence of medical or surgical conditions which could prevent the subject from complying with study procedures.
2. Serum alanine transaminase (ALT) levels above 2x upper limit of normal (ULN) or total bilirubin > 1.3x ULN
3. Serum creatinine levels above 1.5x upper limit of normal
4. Evidence of QT prolongation on electrocardiogram (ECG) QTc (Rate adjusted QT interval) > 450ms (men) or 460ms (women)
5. Pregnant women or female subjects who are unwilling to use a suitable contraceptive method for the duration of the study (IUD or contraceptive implant)
6. Likely to be poorly adherent based on clinician's medical judgement
7. Known to be current injection drug user

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Number of adverse events categorised by body system | 30 days
  The number of adverse events will be tabulated by body system. All safety parameters will be listed by cohort, subject and visit/time and summarized by treatment and visit/time. No formal statistical hypotheses of the safety or tolerability are to be tested.
Percentage of participants with adverse events categorised by body system | 30 days
  The incidence of adverse events will be tabulated by body system. All safety parameters will be listed by cohort, subject and visit/time and summarized by treatment and visit/time. No formal statistical hypotheses of the safety or tolerability are to be tested.
Peak Concentration (CMax) of remdesivir in peripheral blood mononuclear cells (PBMCs) and Plasma | last measurable time-point (24 hours)
  maximum plasma and intracellular concentration [Cmax] of remdesivir with or without co-administration of antiretroviral drugs.
Time to maximum concentration (TMax) of remdesivir in peripheral blood mononuclear cells (PBMCs) and Plasma | last measurable time-point (24 hours)
  Time to maximum concentration of remdesivir in plasma and PBMCs with or without co-administration of antiretroviral therapy
Terminal elimination half-life of remdesivir in plasma and PBMCs | 24 hours
  terminal elimination half life of remdesivir in peripheral blood mononuclear cells (PBMCs) and Plasma with or without co-administration of antiretroviral therapy.
Area under concentration-time curve (AUC) of remdesivir | last measurable time-point (24 hours)
  Area under concentration-time curve of remdesivir in peripheral blood mononuclear cells (PBMCs) and Plasma with or without co-administration of antiretroviral therapy.

SECONDARY OUTCOMES:
Geometric mean ratio and 90% confidence intervals of remdesivir CMax with and without antiretroviral therapy. | 24 hours
  CMax of remdesivir in plasma and PBMCS will be compared with and without antiretroviral therapy.
Geometric mean ratio and 90% confidence intervals of remdesivir TMax with and without antiretroviral therapy. | 24 hours
  TMax of remdesivir in plasma and PBMCS will be compared with and without antiretroviral therapy.
Geometric mean ratio and 90% confidence intervals of remdesivir terminal elimination half-life with and without antiretroviral therapy. | 24 hours
  t 1/2 of remdesivir in plasma and PBMCS will be compared with and without antiretroviral therapy.
Geometric mean ratio and 90% confidence intervals of remdesivir area under concentration-time curve, with and without antiretroviral therapy. | 24 hours
  AUC (0-t) of remdesivir in plasma and PBMCS will be compared with and without antiretroviral therapy. t is the last measurable time-point

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed J Lamorde, PhD, Principal Investigator — Infectious Diseases Institute, Uganda
Locations (1):
- Infectious Diseases Institute, Kampala, Uganda

REFERENCES:
- [Derived] Walimbwa SI, Kaboggoza JP, Waitt C, Byakika-Kibwika P, D'Avolio A, Lamorde M. An open-label, randomized, single intravenous dosing study to investigate the effect of fixed-dose combinations of tenofovir/lamivudine or atazanavir/ritonavir on the pharmacokinetics of remdesivir in Ugandan healthy volunteers (RemTLAR). Trials. 2021 Nov 23;22(1):831. doi: 10.1186/s13063-021-05752-1. PMID 34814933